CLINICAL TRIAL: NCT05255705
Title: Barts Revascularisation Registry - To Understand the Characteristics, Time-trends and Outcomes in Patients With Coronary Artery Disease at Barts Heart Centre
Brief Title: Barts Revascularisation Registry
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE ID: 142567
Record Dates: First submitted 2022-01-18; First posted 2022-02-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction; Stable Angina
MeSH Terms: conditions — Myocardial Infarction; Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing Revascularisation at Barts Heart Centre: This study aims to assess, in a real-world setting, the safety, efficacy and feasibility of further investigations in patients with coronary artery disease undergoing revascularisation.
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — Observation only

SUMMARY:
Despite the year-on-year decrease, coronary artery disease (CAD) still remains one of the leading cause of mortality worldwide. With advances in technology and our understanding of cardiac disease, we can now treat CAD using minimally invasive interventional techniques. This has revolutionised treatment for and improved the lives of many patients with CAD. Although trials have assessed various therapeutic strategies in various populations, real-world evidence of intervention and medical treatment among patients with CAD is increasingly recognised as an important part of providing safety and efficacy data and improving the care we provide.

This data will add to that literature by assessing the characteristics and outcomes of patients with CAD. It will also identify and characterise predictors of outcomes, improve risk stratification and diagnostic evaluation.

DETAILED DESCRIPTION:
The collection of data to describe the nationwide practice of percutaneous coronary intervention (PCI) in the UK started with the inception of the British Cardiovascular Intervention Society (BCIS) in 1988. From 1988 to 1991 annual surveys of PCI activity were published in the British Heart Journal. Annual reports from 1992 onwards are available for download from the society's website (http://www.bcis.org.uk), and summaries of some of the key data have been published as reports for distribution to participating hospitals and networks. The initial data collection process was essentially a descriptive survey of activity. Over time the process has evolved becoming more sophisticated with electronic methods for data collection developed by the Central Cardiac Audit Database (CCAD) group. The methods were tested in 1996 as a pilot in selected hospitals, and full UK-wide participation in the electronic collection of PCI data was achieved by 2005.

The proposed study includes one of the largest coronary interventional and surgical programmes in the UK at Europe's largest cardiac centre (BHC). This has allowed us to accumulate a large number of patients in just over 4 years. All patients undergoing PCI and CABG are included in this study using a clinical database. The database is password-protected and includes demographic, clinical and outcome data.

The database includes patients with simple to complex CAD. We will use this database to test several hypothesis including but not limited to investigating characteristics of patients treated, complications of interventional treatment and outcomes of patients. This research will add substantially to the literature by providing real-world data from a leading coronary centre.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will not be sought for, as patients are automatically included onto a database that we will use for research purposes.
* No children will be included in this study.
* Vulnerable adults or those unable to give consent will be included in the study as well if they are referred to the Interventional Cardiology team.
* Both male and female patients ≥16 years of age will be included
* All patients will have had an angiogram at BHC.
* Any patient who has undergone revascularisation.

Exclusion Criteria:

• Patients <16 years will not be included in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include all patients admitted to or reviewed at Barts Heart Centre (St. Bartholomew's Hospital) who undergo revascularisation. These patients range from young adults to the elderly and will include any patient ≥16 years of age. Patients who are followed up with and without any intervention (i.e. both medically managed patients as well as patients undergoing intervention) are equally as important and therefore we shall include both groups of patients.
  Patients will be included from referrals made by other clinicians either as in or outpatients. All these patients have their clinical data captured on a database or hospital based clinical programme.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year
  Assessment of Mortality
Re-admission rates post Revascularisation | 1 year
  Re-admission
MACE post Revascularisation | 1 year
  MACE

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No